CLINICAL TRIAL: NCT02422706
Title: Study of Nitazoxanide (NTZ) Based New Therapeutic Regimens for Helicobacter Pylori
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sherief Abd-Elsalam (Other)
Collaborators: Tanta University (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, Tanta university, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HELICOBACTER NEW TREATMENT
Record Dates: First submitted 2015-04-13; First posted 2015-04-21 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Helicobacter-associated Gastritis
MeSH Terms: interventions — nitazoxanide; Metronidazole; Omeprazole; Clarithromycin; Levofloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: blinding was applied by using consecutively numbered envelopes that contained the treatment assignments
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- group I (Active Comparator): Metronidazole(MTZ) 500mg twice daily ,Omeprazole 20 mg twice daily as (Proton Pump Inhibitor (PPI)& Clarithromycin 500 mg twice daily .for 14 days .
  40 patients
  Interventions: Drug: Metronidazole(MTZ); Drug: Omeprazole; Drug: Clarithromycin
- Group II (Experimental): Nitazoxanide(NTZ)500 mg twice daily ,PPI 20 mg twice daily & Clarithromycin 500 mg twice daily for 14 days.
  40 patients.
  Interventions: Drug: Nitazoxanide; Drug: Clarithromycin
- Group III (Experimental): Levofloxacin 250 mg once daily,Omeprazole 40mg once daily(PPI),Nitazoxanide (NTZ) 500mg twice daily & Doxicycline 100 mg once daily (LOND).
  40 patients
  Interventions: Drug: Nitazoxanide; Drug: Omeprazole; Drug: Levofloxacin; Drug: Doxicycline

INTERVENTIONS:
Drug: Nitazoxanide — Nitazoxanide based treatment regimens as a new treatment regimens for helicobacter pylori infection
  Other Names: Alenia,parazoxanide,Nitclean
  Arms: Group II; Group III
Drug: Metronidazole(MTZ) — Metronidazole 500 mg twice daily
  Other Names: Flagyl
  Arms: group I
Drug: Omeprazole — Omeprazole 20 twice daily
  Other Names: Omepak. Napizole
  Arms: Group III; group I
Drug: Clarithromycin — KLacid twice daily
  Other Names: KLacid
  Arms: Group II; group I
Drug: Levofloxacin — Tavanic. Tavacin
  Other Names: Levofloxacin once daily
  Arms: Group III
Drug: Doxicycline — Vibramycin 100 mg twice daily
  Other Names: vibramycin. Doxymycin
  Arms: Group III

SUMMARY:
Current Helicobacter Pylori infection preferred treatment involves; proton pump inhibitor (PPI)-based triple or qudrable regimens. Omeprazole, Amoxicillin, and Clarithromycin is one of a global standard care for confirmed H.pylori infection . Metronidazole (MTZ) is used instead of Amoxicillin or Clarithromycin in cases of allergy or resistance .

However, a recent study based on the Maastricht III guidelines, indicated that treatment with a PPI-based triple regimen as first-line therapy will fail in ~30% of patients on an intention-to-treat (ITT) basis, and will fail in ~ 50 % of patients who treated with PPI-based triple regimen with Metronidazole. This treatment resistance is also an issue warranting the investigation of other agents. Helicobacter pylori infection has become increasingly resistant to traditional first-line treatment regimens because of emerging antibiotic resistance coupled with poor patient compliance with completing the treatment course that decrease H. pylori eradication rates. So there is a considerable interest in evaluating new antibiotic combinations and regimens .

DETAILED DESCRIPTION:
Helicobacter pylori (H.pylori) is a small, Gram-negative spirochete inhabiting the mucous layer overlying the gastric epithelial cells in humans. It is the most common prevalent chronic human bacterial infection and the most common cause of gastritis worldwide;. Furthermore, according to the World Health Organization, HP is classified as a type 1 carcinogen and is the primary cause of peptic ulcer disease, gastric carcinoma, and mucosa-associated lymphoid tissue lymphomas .

Current Helicobacter Pylori infection preferred treatment involves; proton pump inhibitor (PPI)-based triple or qudrable regimens.Omeprazole,Amoxicillin &Clarithromycin is one of a global standard care for confirmed H.pylori infection .Metronidazole (MTZ) is used instead of Amoxicillin or Clarithromycin in cases of allergy or resistance .

However, a study by Rokkas , et al., 2008 based on the Maastricht III guidelines, indicated that treatment with a PPI-based triple regimen as first-line therapy will fail in ~30% of patients on an intention-to-treat (ITT) basis,and will fail in ~ 50 % of patients who treated with PPI-based triple regimen with Metronidazole.This treatment resistance is also an issue warranting the investigation of other agents . Helicobacter pylori infection has become increasingly resistant to traditional first-line treatment regimens because of emerging antibiotic resistance coupled with poor patient compliance with completing the treatment course that decrease H. pylori eradication rates .So there is a considerable interest in evaluating new antibiotic combinations and regimens.

Nitazoxanide (NTZ) is an antibiotic with microbiological characteristics similar to those of Metronidazole which was sittled as a therapy for intestinal protozoa and helminthic infection,and was studied as an additional therapy with Peg Interferon and Ribavirin for chronic hepatitis C virus (HCV) .

In the last few years Nitazoxanide was evaluated as a single agent therapy for H. Pylori infection showing controversed results.. However (NTZ) based regimens were recently studied showing interesting results without the apparent problem of resistance as Metronidazole with nearby cost.Moreover ;Levofloxacin,PPI,NTZ&Doxycycline (LOAD) regimen with very good results in H.pylori infection ~90% cure rate..But uptil now there are no actual similar reported trials in Egypt.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with dyspeptic symptoms undergoing upper Gasto-intestinal tract (GIT) endoscopy selecting HP infected patients to be recruited for the study.
* Patients must have had Helicobacter Pylori - induced disease confirmed by endoscopy and HP monoclonal stool antigen.

Exclusion Criteria:

1. Previous gastric or duedenal operations or malignancy.
2. Active GIT bleeding.
3. Pregnancy.
4. Previous treatment for HP.
5. Current use of Antiacids ( proton pump inhibitor ( PPI ), H2 receptor antagonist) , anticoagulant, or recent use of antibiotics (within 6 weeks).
6. Allergy to any medication included in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with proven eradication of helicobacter | 6 weeks
  Number of patients with proven eradication of helicobacter after 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mona AH Shehata, Prof, Study Chair — liver dis dept; Sherief Abd-Elsalam, Consultant, Study Director — Division of Gastroenterology and Hepatology- Tanta; Raghda Talaat, Prof, Study Chair — Microbiology; Huda Elmesseri, Specialist, Study Chair — liver diseases dept.-Elmahalla hospital
Locations (1):
- Tanta university hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shehata MA, Talaat R, Soliman S, Elmesseri H, Soliman S, Abd-Elsalam S. Randomized controlled study of a novel triple nitazoxanide (NTZ)-containing therapeutic regimen versus the traditional regimen for eradication of Helicobacter pylori infection. Helicobacter. 2017 Oct;22(5). doi: 10.1111/hel.12395. Epub 2017 May 19. PMID 28524341